CLINICAL TRIAL: NCT01473641
Title: Nexplanon Observational Risk Assessment Study (NORA)
Acronym: NORA
Status: Completed | Type: Observational
Sponsor: Center for Epidemiology and Health Research, Germany (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Klaas Heinemann, MD, PhD, Principal Investigator, Center for Epidemiology and Health Research, Germany
Other Study IDs: ZEG2011_03
Record Dates: First submitted 2011-11-15; First posted 2011-11-17 (Estimated); Last update posted 2019-11-07 (Actual); Status verified 2019-11

CONDITIONS: Contraception
Keywords: Etonogestrel; Contraceptive implant; Safety

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- New users of Nexplanon

SUMMARY:
This study characterises the frequency of specific insertion-, localization- and removal-related events and clinically significant consequences thereof among Nexplanon users in the US during routine clinical use.

DETAILED DESCRIPTION:
Nexplanon is a subdermal contraceptive implant containing the progestogen etonogestrel. It provides contraceptive protection for three years. In addition to the progestogen, Nexplanon contains barium sulfate and a Next Generation Implanon Applicator (NGIA). Nexplanon was developed to further facilitate correct insertion of the implant by using the NGIA, and to extend the diagnostic modalities for localization of the implant by making it radiopaque and visible via X-ray imaging and X-ray Computerized Tomography (CT).

A large, descriptive, prospective, non-interventional, observational cohort study is planned to follow a cohort of new users of the contraceptive implant Nexplanon. Women will be recruited through health care professionals who have completed the Nexplanon Clinical Training Program. Baseline and follow-up information will be collected via a self-administered questionnaire. Data analysis will include characterizing the frequency of specific insertion-, localization- and removal-related events via point-estimates of the event rate as well as 95% confidence intervals. The impact of potential prognostic factors will be analyzed using multivariate regression models and/or stratified analyses.

ELIGIBILITY:
Inclusion Criteria:

* Women prescribed a new Nexplanon implant
* Women who are capable of understanding the major aspects of the study and can complete the self-administered questionnaire in English

Exclusion Criteria:

* Women who are not willing to sign the informed consent form

Min Age: 12 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Women using the contraceptive implant Nexplanon
Sampling Method: Non-Probability Sample
Enrollment: 7364 (Actual)
Dates: Start 2011-11; Primary Completion 2017-10-31 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
Insertion-, localization- and removal-related events | Within 42 months after insertion
  Incorrect insertion (i.e. unrecognized non-insertion, partial insertion, deep insertion); palpability of the implant at insertion and removal; localization of a non-palpable implant; difficult removals; pregnancy due to unrecognized non-insertion of the implant; injury to neurovascular structures in the arm; hospitalization and/or surgical procedures for localization and/or removal.

SECONDARY OUTCOMES:
Pregnancy | Within 42 months after insertion
  Pre-treatment, in-treatment, post-treatment and non-insertion pregnancies.
Pregnancy outcomes | Within 42 months after insertion
  Pregnancy outcomes in pregnancies where fetal exposure to etonogestrel may have taken place.
Reasons for (premature) discontinuation of Nexplanon | Within 42 months after insertion
  The reason(s) the patient had the implant removed.
Baseline characteristics of Nexplanon users | Within 42 months after insertion
  Baseline characteristics (including contraceptive history, medical history, gynecological history and socio-demongraphic details).

CONTACTS AND LOCATIONS:
Overall Officials: Klaas Heinemann, MD, MBA, PhD, Principal Investigator — Center for Epidemiology and Health Research, Berlin, Germany
Locations (1):
- Center for Epidemiology and Health Research, Berlin, Germany

REFERENCES:
- [Result] Reed S, Do Minh T, Lange JA, Koro C, Fox M, Heinemann K. Real world data on Nexplanon(R) procedure-related events: final results from the Nexplanon Observational Risk Assessment study (NORA). Contraception. 2019 Jul;100(1):31-36. doi: 10.1016/j.contraception.2019.03.052. Epub 2019 Apr 10. PMID 30980829

DOCUMENTS (2):
  • Study Protocol (2011-07-15): https://cdn.clinicaltrials.gov/large-docs/41/NCT01473641/Prot_000.pdf
  • Statistical Analysis Plan (2011-08-01): https://cdn.clinicaltrials.gov/large-docs/41/NCT01473641/SAP_001.pdf